CLINICAL TRIAL: NCT07184437
Title: A Clinical Investigation of MINIVISC® PLUS 14 mg/ml Fermented Ophthalmic Viscosurgical Device (OVD-F), Used for Cataract Surgery and Implantation of Intraocular Lenses, Glaucoma Surgery, Anterior Segment Surgery and Corneal Transplantation (CGAC)
Acronym: Minivisc01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bohus Biotech AB (Industry)
Collaborators: Key2Compliance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-23-10-044394
Record Dates: First submitted 2024-08-06; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cataract
Keywords: Cataract surgery; Implantation of intraocular lenses; Glaucoma surgery; Anterior segment surgery; Corneal transplantation
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: In Phase A, eligible subjects will undergo surgery on one or both eyes. In case of both eye surgery, subjects will receive the IMD (MINIVISC®PLUS 14 mg/ml) in one eye and the control OVD (Healon GV® PRO 18 mg/ml OVD) in the other eye. In case of one eye surgery, MINIVISC® PLUS 14 mg/ml OR Healon GV® PRO 18 mg/ml will be randomly assigned to the eye.
  In Phase B, eligible subjects will undergo surgery on one eye. The subjects will receive the IMD (MINIVISC®PLUS 14 mg/ml OVD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase A (Active Comparator): In Phase A, eligible subjects will undergo surgery on one or both eyes. In case of both eye surgery, subjects will receive the IMD (MINIVISC®PLUS 14 mg/ml) in one eye and the control OVD (Healon GV® PRO 18 mg/ml OVD) in the other eye. OVDs will be randomly assigned by investigator to each eye to reach an as even as possible distribution of the IMD and comparator. In case of one eye surgery, MINIVISC® PLUS 14 mg/ml OR Healon GV® PRO 18 mg/ml will be randomly assigned to the eye. Healon GV® PRO 18 mg/ml OVD is a legally marketed alternative with similar indications for use and similar properties as the MINIVISC®PLUS 14 mg/ml OVD.
  Interventions: Device: OVD-F device Minivisc®PLUS 14 mg/ml
- Phase B (Other): In the Phase B, eligible subjects will undergo surgery on one eye. The subjects will receive the IMD (MINIVISC®PLUS 14 mg/ml OVD).
  Interventions: Device: OVD-F device Minivisc®PLUS 14 mg/ml

INTERVENTIONS:
Device: OVD-F device Minivisc®PLUS 14 mg/ml — MINIVISC® PLUS 14 mg/ml is intended to protect, lubricate and support delicate ophthalmic cells or tissues, to assist in maintaining intraocular space and to enhance visualization during surgery.

SUMMARY:
A clinical investigation to confirm the clinical safety and performance of OVD-F device MINIVISC® PLUS 1.4 % for cataract surgery and implantation of intraocular lenses, glaucoma surgery, anterior segment surgery and corneal transplantation.

DETAILED DESCRIPTION:
The investigation will include two phases, Phase A and Phase B. The duration of the patient follow-up in Phase A is 90 days, in Phase B - 7 days, alternatively 30 days, depending on intraocular pressure, during which the safety and performance of the IMD will be assessed. AEs will be followed up until resolution or the follow-up assessment, whichever comes first, or according to the judgement of the PI or authorized designee.

In Phase A, eligible subjects will undergo surgery on one or both eyes. In case of both eye surgery, subjects will receive the IMD (MINIVISC®PLUS 14 mg/ml) in one eye and the control OVD (Healon GV® PRO 18 mg/ml OVD) in the other eye. OVDs will be randomly assigned by investigator to each eye to reach an as even as possible distribution of the IMD and comparator. In case of one eye surgery, MINIVISC® PLUS 14 mg/ml OR Healon GV® PRO 18 mg/ml will be randomly assigned to the eye.

Healon GV® PRO 18 mg/ml OVD is a legally marketed alternative with similar indications for use and similar properties as the MINIVISC®PLUS 14 mg/ml OVD.

In the Phase B, eligible subjects will undergo surgery on one eye. The subjects will receive the IMD (MINIVISC®PLUS 14 mg/ml OVD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, >18 years, in need of ophthalmic surgery for:

   * Cataract
   * Glaucoma surgery
   * Anterior segment trauma or diseases
   * Damaged or diseased cornea
2. Able and willing to give informed consent for participation in the investigation.
3. For the participation in Phase A of the study, patients that need surgery on one or both eyes will be included. For the participation in Phase B of the study, patients that need surgery on one or both eyes will be included but only one eye can be included in the clinical investigation.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Any previous hypersensitivity reaction to any constituent of the IMD.
3. Concurrent participation or participation within 45 days prior to preoperative visit in any other clinical trial.
4. Recent ocular trauma or ocular surgery that is not resolved/stable or may affect clinical outcomes or increase risk to the subject.
5. Ocular hypertension of ≥22 mmHg, after 3 repeated measurements pre-surgery.
6. An endothelial cell count (ECC) lower than 1800 cells/mm2 preoperatively, based on the average of the three cell counts as taken by the Specular Microscope (only in Phase A).
7. Any other condition or treatment making the subject unsuitable for participation in the clinical investigation, as judged by the Principal Investigator, including but not exclusive to diagnosis of wide-angle glaucoma, severe myopia, uveitis, and physical traits such as a small pupil, an extremely shallow anterior chamber, or a compromised endothelial cell function.
8. Employees of the study site or the sponsor directly involved with the conduct of the investigation, or immediate family members of any such individuals.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint is the postoperative intraocular pressure (IOP) | 7 days
  The primary endpoint is the postoperative intraocular pressure (IOP). A patient is defined as a failure if the IOP ≥ 30 mmHg within 7 days post-surgery (Data from Phase A and Phase B pooled, IMD only).

SECONDARY OUTCOMES:
Secondary endpoint is the Postoperative inflammation, as measured by slit-lamp bio-microscopy, and graded using a standard grading system, such as The Standardization of Uveitis Nomenclature (SUN) Working group | +2hours, 7, 30 and 90 days,
  Postoperative inflammation, as measured by slit-lamp bio-microscopy, and graded using a standard grading system, such as The Standardization of Uveitis Nomenclature (SUN) Working group, at the 2-hour post-surgery follow-up, and at the 7-, 30- and 90-days follow-up visits, as applicable according to the investigational design.
Secondary endpoint is the central corneal endothelial cell density (cells/mm2), as measured by Specular Microscope images. | 90 days
  The central corneal endothelial cell density (cells/mm2), as measured by Specular Microscope images, pre-surgery and at 90 days ± 14 days post-surgery (only Phase A).
Secondary endpoint Principal investigator evaluation of adverse events during surgery, and at all follow-up visits. | Assessed during the whole study, in Phase A up to 90 (+/-14d) days, and in Phase B up to 30 (+/- 7d) days.
  Principal investigator evaluation of adverse events during surgery, and at all follow-up visits, as applicable according to the investigational design.
Secondary endpoint is Investigator/surgeon evaluation of IMD performance through ratings of a number of performance related criteria | Assessed by surgeon after surgery +2h
  Investigator/surgeon evaluation of IMD performance, immediately post-surgery, through ratings of a number of performance related criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Johansson, MD, Principal Investigator — Opthalmic Clinic University Hospital Linköping
Locations (6):
- UZ Leuven, Leuven, Belgium
- Sweden (5):
  - Eye Clinic Falu Hosptal, Falun, Dalarna County
  - Ögonläkargruppen Odenplan, Stockholm, Stockholm County
  - Optalmica Eye Clinic, Stockholm, Stockholm County
  - Optalmic Clinic Uddevalla Hospital, Uddevalla, Västra Götaland County
  - Opthalmic Clinic University Hospital Linköping, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No